CLINICAL TRIAL: NCT06149065
Title: Factors Associated With the Acne Severity Among Transmen Population: a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 2124
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Acne; Transgenderism
Keywords: Diet, Female-to-male transgender, Masculinizing hormone therapy, Risk factors
MeSH Terms: conditions — Acne Vulgaris; Transsexualism | interventions — Testosterone; Demography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 17 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Testosterone — Masculinizing hormone therapy (testosterone) is used in female-to-male transgenders for medical reason.
  Other Names: Demographic data, acne-related clinical risk factors

SUMMARY:
The goal of this observational cross-sectional study is to identify factors associated with severity of acne in Thai transmen receiving masculinizing hormone therapy. The main questions it aims to answer are:

* What are the factors associated with severity of acne in transmen?
* Does masculinizing hormone therapy associate with the severity of acne in transmen? Participants will be asked to complete an online questionnaire and allow to take pictures of their face for acne assessment purpose.

ELIGIBILITY:
Inclusion Criteria:

* Transmen who visited the Gender Variation (GenV) Clinic of Ramathibodi Hospital
* Transmen who received masculinizing hormone therapy (testosterone)
* Transmen who completed an online questionnaire and intentional submit their facial photographs

Exclusion Criteria:

* Refusal to participate
* Incomplete questionnaire
* Missing photos
* Diagnosis of any disorders of sexual differentiation which may have peculiar hormonal effect

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender male (also: trans man, female-to-male, transgender male): this refers to individuals assigned female at birth but who identify and live as men.
Study Population: All transmen who visited the Gender Variation (GenV) Clinic (outpatient clinic) of Ramathibodi Hospital
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
The severity of acne | 1 day (At the time of answering an online questionnaire)
  Investigator Global Assessment (IGA) scale for acne

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Dermatology, Department of Internal Medicine, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided